CLINICAL TRIAL: NCT06641505
Title: Feasibility of Deep Inspiratory Internal Jugular Vein Variability in Guiding Preoperative Fluid Replacement：A Prospective, Randomized Controlled Study
Brief Title: Feasibility of Deep Inspiratory Internal Jugular Vein Variability in Guiding Preoperative Fluid Replacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, Principal investigator, Affiliated Hospital of Jiaxing University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-KY-520
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-08

CONDITIONS: Hemodynamic
Keywords: Internal jugular vein; propofol; hemodynamic; hypotension; fluid replacement
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guiding rehydration group (Experimental): According to the 421 fluid replacement principle, preoperative fluid replacement is performed
  Interventions: Behavioral: Guiding rehydration
- Conventional rehydration group (Active Comparator): rehydrated within 15 minutes according to 0.2ml/kg/min.
  Interventions: Behavioral: Guiding rehydration

INTERVENTIONS:
Behavioral: Guiding rehydration — Preoperative fluid rehydration was performed according to 421 fluid rehydration principles

SUMMARY:
Compare the incidence of hypotension during the propofol-induced period between the internal jugular vein variability-guided fluid infusion group and the conventional fluid infusion group through a fluid infusion experiment before anesthesia induction, so as to evaluate the feasibility of using the internal jugular vein variability under deep inspiration to guide preoperative fluid infusion.

DETAILED DESCRIPTION:
Ultrasound records at least one quiet breathing cycle and one deep inhalation cycle to calculate IJVV Propofol was infused target-controlled at 4 μg/ml, and changes in arterial blood pressure within 3 minutes of propofol induction were observed.

Plan to conduct a prospective randomized controlled study to compare the incidence of hypotension during the propofol-induced period between the internal jugular vein variability-guided fluid infusion group and the conventional fluid infusion group through a fluid infusion experiment before anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* age over 60 years； American Society of Anesthesiology (ASA) status Ⅱ-Ⅲ； Surgery with radial artery puncture； Propofol induction；

Exclusion Criteria:

* BMI≥30kg/m2； People with short necks； Previous hypotension (systolic blood pressure <90mmHg or mean arterial pressure<65mmHg)； Previous poorly controlled hypertension； Cardiac insufficiency , EF value<50%； Upper limb deep vein thrombosis； History of radiotherapy or neck surgery； Inability to maintain a supine position for necessary measurements； Mechanical ventilation status or inability to take deep breaths patients； gastrointestinal surgery； Patients allergic to propofol； Restricted fluid intake；

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of a 20% drop in blood pressure after propofol induction | 1 year
  The incidence of a 20% drop in blood pressure after propofol induction

CONTACTS AND LOCATIONS:
Overall Officials: Qinghe Zhou, Principal Investigator — Affiliated Hospital of Jiaxing University
Locations (1):
- Affiliated Hospital of University, Jiaxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei XL, Xi YZ, Xie L, Li ZP, Tang HL, Zhou QH. Effects of liquid resuscitation guided by internal jugular vein variability during deep inhalation on preventing propofol-induced hypotension in elderly patients. BMC Anesthesiol. 2025 Jul 17;25(1):350. doi: 10.1186/s12871-025-03227-3. PMID 40676549